CLINICAL TRIAL: NCT00982852
Title: Intravascular Ultrasound Derived Virtual Histology and Intracoronary Serum Markers of Inflammation in Patients Referred for Percutaneous Coronary Intervention.
Brief Title: Intravascular Ultrasound Derived Virtual Histology and Intracoronary Serum Markers of Inflammation
Status: Terminated | Type: Observational
Why Stopped: Lack of funding
Sponsor: Quinn Capers (Other)
Responsible Party: Sponsor-Investigator, Quinn Capers, Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2008H0112
Record Dates: First submitted 2009-01-26; First posted 2009-09-23 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Myocardial Infarction; Heart Failure; Angina
Keywords: Angioplasty; Coronary Vessels; Heart Disease; Cardiology; Atherosclerosis; Catheterization
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Myocardial Infarction; Heart Failure; Angina Pectoris; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood that is collected will be analyzed for markers of inflammation or irritation in the blood (c-reactive protein, myeloperoxidase, Monocyte chemotactic protein-1), as well and a gene called Matrix Metallopeptidase 3, which is believe to influence the progression of plaque on the walls of arteries and the progression of coronary artery disease.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute: Patients in acute need for angioplasty or left heart catheterization.
- Chronic or non-acute: Patients will planned angioplasty or left heart catheterization.

SUMMARY:
Patients enrolled will need treated with an IVUS- VH (intravascular ultrasound-derived virtual histology) which is an arterial stent procedure, that involves threading a tiny wire into the artery, followed by a balloon, a stent, or other device to treat a blocked artery, and often (though not always), a special ultrasound catheter to take pictures of the inside of the artery.

Participants in the study, will have an additional procedure performed: a tiny tube will be advanced into the heart artery to collect a blood sample for research purposes, and a blood sample will be collected from the femoral (thigh) artery through the tube that will be placed there as a standard part of having this procedure.

The blood that is collected will be analyzed for markers of inflammation or irritation in the blood (c-reactive protein, myeloperoxidase, Monocyte chemotactic protein-1), as well and a gene called Matrix Metallopeptidase 3, which is believe to influence the progression of plaque on the walls of arteries and the progression of coronary artery disease. .

DETAILED DESCRIPTION:
Patients that have severe blockage in one of the arteries that provides blood flow to your heart will be enrolled into the research study. Most of the procedures in the study standard care used by cardiologists when treating blocked arteries. Patients enrolled will need treated with an IVUS- VH (intravascular ultrasound-derived virtual histology) which is an arterial stent procedure, that involves threading a tiny wire into the artery, followed by a balloon, a stent, or other device to treat a blocked artery, and often (though not always), a special ultrasound catheter to take pictures of the inside of the artery. We will collect all the data from the above stated standard medical care procedure.

Participants in the study, will have an additional procedure performed: a tiny tube will be advanced into the heart artery to collect a blood sample for research purposes, and a blood sample will be collected from the femoral (thigh) artery through the tube that will be placed there as a standard part of having this procedure.

The blood that is collected will be analyzed for markers of inflammation or irritation in the blood (c-reactive protein, myeloperoxidase, Monocyte chemotactic protein-1), as well and a gene called Matrix Metallopeptidase 3, which is believe to influence the progression of plaque on the walls of arteries and the progression of coronary artery disease. .

Finally, after discharged from the hospital, the research nurses will call you at home to ask you questions about how you are doing for approximately 5-10 minutes. Telephone follow-up will occur at one month, six months, 12 months, 18 months, 24 months, and 36 months.

ELIGIBILITY:
Inclusion Criteria:

* In- or out-patients admitted to IPR or hospital floor for left heart catheterization or scheduled angioplasty
* 18 years or older
* Able to provide informed consent

Exclusion Criteria:

* Patients who are pregnant or lactating
* Inability to provide informed consent
* Patients undergoing heart catheterization for who open heart surgery is planned
* Anticipate being unavailable for telephone follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of angioplasty or left heart catheterization
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Occurrence or absence of adverse cardiovascular outcomes up to 36 months after PCI | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Quinn Capers IV, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States